CLINICAL TRIAL: NCT02889081
Title: Maternal Key Nutritional Factors and Offspring's Atopic Dermatitis
Brief Title: Maternal Key Nutritional Factors and Offspring's Atopic Dermatitis (MKNFOAD)
Acronym: MKNFOAD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Minhang Maternal and Children Health Care Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AD2016-2018
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
Keywords: birth cohort; prenatal; skin barrier; atopic dermatitis; key nutritional factors
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Maternal venous blood and offspring's cord blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- infants from birth cohort with AD: maternal biological folate level and maternal biological vitamin D level and offspring's incidence of suffering from atopic dermatitis
  Interventions: Other: maternal biological folate level; Other: maternal biological Vitamin D level
- infants from birth cohort without AD: maternal biological folate level and maternal biological vitamin D level and offspring's incidence of not suffering from atopic dermatitis
  Interventions: Other: maternal biological folate level; Other: maternal biological Vitamin D level

INTERVENTIONS:
Other: maternal biological folate level — supplementation status and serum level
Other: maternal biological Vitamin D level — supplementation status and serum level

SUMMARY:
The study is a prospective birth cohort study and the purpose is to describe the status of maternal key nutrients(eg. folate and vitamin D) supplementation among pregnancies at early gestation in Shanghai, to find out the association between the level of serum key nutrients and atopic dermatitis (AD) in offsprings during 6 months.

DETAILED DESCRIPTION:
This study based on Shanghai pregnancy population is a prospective birth cohort. The investigators obtain the data of participants' folic acid and vitamin D supplement intake through the questionnaire at 12-14 gestational weeks. And the investigators collect participants' blood samples during gestation to directly detect the biological exposure levels of folate and vitamin D. In the follow-up, skin barrier function is evaluated at time of infant 24-48 hours, 42 days and 6 months. During 6 months from birth, the incidence of AD is investigated on offsprings. This cohort study is aimed to (1) clarify the association between prenatal key nutrients with offspring AD; (2) assess the role of maternal key nutrients in the skin barrier of offsprings. It will be a good evidence for the AD prevention and a meaningful protocol to reduce the incidence of AD by its unique design.Univariate and multivariate association analyses will be performed to identify risk factors to AD by using multivariate logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Mother plans to proceed prenatal care and delivery in Minhang Maternal and Children Health Care Hospital
* Offspring plans to stay in Shanghai until 6 months and proceed follow-up in Children's Hospital of Fudan University

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregancies at early gestation and offspring from Minhang Maternal and Children Health Care Hospital in Shanghai from June 2016
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Infant atopic dermatitis | incident of AD during 6 months after birth, diagnosis confirmed based on disease history till 12 months
  Disease diagnosis according to the criteria of Williams

SECONDARY OUTCOMES:
Maternal RBC folate level | 12-14 gestational weeks
  Whole blood sample collected will be used for evaluation
Maternal serum vitamin D level | 12-14 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum vitamin D level | 22-26 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum vitamin D level | 34-36 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum folate level | 12-14 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum folate level | 22-26 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum folate level | 34-36 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal folic acid supplement intake | 12-14 gestational weeks
  Questionnaire survey will be used to obtain the data of maternal supplement intake
Maternal vitamin D supplement intake | 12-14 gestational weeks
  Questionnaire survey will be used to obtain the data of maternal supplement intake
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 24-48 hours
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 42 days old
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Transepidermal Water Loss, TEWL） | infant 6 months old
  TEWL will be evaluated by the device of Multi Probe Adapter 4.
Infant atopic dermatitis incidence by 1year old | from birth , to 12months old
  Disease diagnosis according to the criteria of Williams
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 24-48 hours
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 42 days old
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (Stratum corneum hydration, SCH) | infant 6 months old
  SCH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 24-48 hours
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 42 days old
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (skin surface pH) | infant 6 months old
  Skin pH will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 24-48 hours
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 42 days old
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Infant skin barrier function (sebum content) | infant 6 months old
  Sebum content will be evaluated by the device of Multi Probe Adapter 4.
Maternal serum Vitamin E level | 12-14 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Maternal serum Vitamin A level | 12-14 gestational weeks
  Serum sample collected at different trimesters will be used for evaluation
Child atopic dermatitis from 1 year old to 2 years old | from 1 year old to 2 years old
  Disease diagnosis according to the criteria of Williams
Child atopic dermatitis from 2 years old to 5 years old | from 2 years old to 5 years old
  Disease diagnosis according to the criteria of Williams

CONTACTS AND LOCATIONS:
Overall Officials: Guoying Huang, MD,PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wegienka G, Havstad S, Zoratti EM, Kim H, Ownby DR, Johnson CC. Association between vitamin D levels and allergy-related outcomes vary by race and other factors. J Allergy Clin Immunol. 2015 Nov;136(5):1309-14.e1-4. doi: 10.1016/j.jaci.2015.04.017. Epub 2015 Jun 12. PMID 26078105
- [Result] Kiefte-de Jong JC, Timmermans S, Jaddoe VW, Hofman A, Tiemeier H, Steegers EA, de Jongste JC, Moll HA. High circulating folate and vitamin B-12 concentrations in women during pregnancy are associated with increased prevalence of atopic dermatitis in their offspring. J Nutr. 2012 Apr;142(4):731-8. doi: 10.3945/jn.111.154948. Epub 2012 Mar 7. PMID 22399526
- [Result] Kelleher M, Dunn-Galvin A, Hourihane JO, Murray D, Campbell LE, McLean WHI, Irvine AD. Skin barrier dysfunction measured by transepidermal water loss at 2 days and 2 months predates and predicts atopic dermatitis at 1 year. J Allergy Clin Immunol. 2015 Apr;135(4):930-935.e1. doi: 10.1016/j.jaci.2014.12.013. Epub 2015 Jan 22. PMID 25618747 (Retraction: PMID 33832697 J Allergy Clin Immunol. 2021 Apr;147(4):1526)